CLINICAL TRIAL: NCT05327894
Title: Interfant-21 International Collaborative Treatment Protocol for Infants Under One Year With KMT2A-rearranged Acute Lymphoblastic Leukemia or Mixed Phenotype Acute Leukemia.
Brief Title: Interfant-21 Treatment Protocol for Infants Under 1 Year With KMT2A-rearranged ALL or Mixed Phenotype Acute Leukemia
Acronym: Interfant-21
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: University of Milano Bicocca (Other); Amgen Europe B.V (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-000213-16
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-07

CONDITIONS: Acute Lymphoblastic Leukemia; Mixed Phenotype Acute Leukemia
Keywords: infant under one year; KMT2A-wildtype
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — blinatumomab

STUDY DESIGN:
Intervention Model Description: Definition: Provide details about the Interventional Study Model. Limit: 1000 characters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medium Risk (MR) (Other): Subject is defined as MR if > 6months of age at diagnosis, OR < 6 months of age with White Blood cell Count (WBC) < 300 at diagnosis and good prednisone response. Subject gets 1st cycle of blinatumomab. If MRD is >0.01%, after 1st cycle of blinatumomab, subject will be allocated to HR treatment from that phase, and will be eligible for HSCT. If MRD is undetectable or < 0.01% after the 1st cycle of blinatumomab (TP2) patient will be eligible for replacement of MARMA by 2nd cycle of blinatumomab after receipt of lymphoid style consolidation (Protocol IB) or of myeloid style consolidation (ADE/MAE).
  Interventions: Drug: Blinatumomab
- High risk (HR) (Other): Subject is defined as HR if < 6 months of age with WBC > 300 at diagnosis OR poor prednisone response. Also MR patients with end of induction MRD ≥ 1%, or MRD > 0.01% after the 1st cycle of blinatumomab, will be allocated to HR treatment. Subject gets 1 cycle of blinatumomab.
  Thereafter patient is eligible for hematopoietic stem cell transplantation (HSCT) with or without experimental therapy in an investigational window.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — 1st cycle: 15 μg/m2/day as a 4 week continuous IV infusion for patients with a M1 marrow. For patients with a M2/M3 marrow a step-dosing strategy is required with a dose of 5 μg/m2/day in week 1 followed by 15 μg/m2/day in weeks 2, 3, and 4.
  Other Names: Cycle 1
Drug: Blinatumomab — 2nd cycle: 15 μg/m2/day as a 4 week continuous iv infusion
  Other Names: Cycle 2
  Arms: Medium Risk (MR)

SUMMARY:
This study is a treatment protocol with blinatumomab for infants under 1 year old who are diagnosed with acute lymphoblastic leukemia with a specific unfavorable genetic alteration. The purpose of the study is to improve the outcome of this disease in infants.

DETAILED DESCRIPTION:
All infants that are eligible for this study and for whom the parents/legal representatives give informed consent will be enrolled in this study. All patients will receive one cycle of blinatumomab on top of the standard treatment backbone after induction therapy. Medium risk patients, that respond well to the 1st cycle will be treated with a 2nd cycle of blinatumomab replacing one chemo course after consolidation therapy. If they do not respond well enough they will be treated according to the current treatment standard. Minimal residual disease will be used to determine the response to blinatumomab. High risk patients will be eligible for allogeneic stem cell transplantation after the first blinatumomab cycle if they are Minimal Residual Disease (MRD) negative (defined as < 0.01%). Also medium risk patients with insufficient MRD response after induction or after the 1st cycle of blinatumomab will be allocated to high risk treatment and will be eligible for allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed B- precursor ALL or B-cell MPAL (single lineage) according to the WHO classification of tumours of haematopoietic and lymphoid tissues (revised 4th edition 2017), with KMT2A-rearrangement.
2. ≤ 365 days of age at the time of diagnosis of ALL.
3. Written informed consent of the parent(s) or other legally authorized guardian of the patient according to local law and regulations.

Exclusion criteria for blinatumomab:

1. KMT2A-wildtype patients.
2. Multilineage MPAL
3. T-ALL.
4. Age > 365 days at the time of diagnosis.
5. Down syndrome.
6. Relapsed ALL.
7. Treatment with systemic corticosteroids (equivalent prednisone >10 mg/m2/day) for more than one week and/or any chemotherapeutic agent in the 4-week interval prior to diagnosis. Patients who received corticosteroids by aerosol are eligible for the study.

If exclusion criteria for blinatumomab are met, the patient should be treated according to the protocol but without blinatumomab.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS). | 5 years
  The primary endpoint is EFS, defined as the time from diagnosis to resistance to induction, relapse, death from any cause or second malignancy (whichever occurs first), or time to last follow-up (censored) for patients without events.

SECONDARY OUTCOMES:
Overall survival | 8 years
  The endpoints for analysis by risk group will be EFS, cumulative incidence (or percentage) of resistance to induction, cumulative incidence of relapse (CIR), death in complete remission (CR) and second malignancy.
Endpoints by risk group | 8 years
  The endpoints for analysis by risk group will be EFS, cumulative incidence (or percentage) of resistance to induction, cumulative incidence of relapse (CIR), death in complete remission (CR) and second malignancy.
Outcome for the entire study cohort and according to risk group | 8 years
  Outcome for the entire study cohort and according to risk group will be evaluated in terms of the protocol specific definition of EFS follows: the time from diagnosis to, resistance to proto-col, relapse, death from any cause or second malignancy (whichever occurs first), or time to last follow-up for patients without events. Cumulative incidence (or percentage) of resistance, CIR, death in CR and second malignancy will also be estimated.
Minimal Residual Disease | 8 years
  MRD response as defined in the protocol and frequencies of MRD levels
CD19 (cluster of differentiation antigen 19) negative relapse | 8 years
  Proportion of CD19 negative relapses in the entire study cohort and according to risk group
Myeloid lineage switches | 8 years
  Proportion of myeloid lineage switches in the entire study cohort and according to risk group
Grade ≥3 adverse event | 8 years
  Proportion of grade ≥3 adverse event (AEs) during the blinatumomab course(s). Proportion of adverse events of special interest (AESIs) and serious adverse events (SAEs) in all protocol phases.
Grade ≥2 cardiac disorders | 5 years
  Proportion of grade ≥2 cardiac disorders at 2 and 5 years after diagnosis
Overall survival after 1st relapse | 8 years
  Overall survival (OS) after first relapse, defined as the time from first relapse to death from any cause, in the entire study cohort and according to risk group

CONTACTS AND LOCATIONS:
Overall Officials: Janine Stutterheim, Dr, Principal Investigator — Princess Maxima Center for Pediatric Oncology in The Netherlands
Locations (112):
- Hospital de Pediatría S.A.M.I.C. "Juan P. Garrahan", Buenos Aires, Argentina
- Australia (9):
  - Australian and New Zealand Children's Haematology/Oncology Group, Clayton, Victoria
  - North Adelaide- Womens and Childrens Hospital, Adelaide
  - Monash Children's Hosptial, Clayton
  - New Lambton Heights- John Hunter Children's Hospital, New Lambton Heights
  - Royal Children's Hospital (Children's Cancer Centre), Parkville
  - Perth Children's Hospital, Perth
  - Queensland Children's Hospital, South Brisbane
  - Sydney Childrens Hospital, Sydney
  - The Childrens Hospital at Westmead, Westmead
- Austria (4):
  - Medical University Of Graz, Graz
  - Medical University Of Innsbruck, Innsbruck
  - Gemeinnutzige Salzburger Landes kliniken Betriebsgesellschaft mbH, Salzburg
  - St. Anna Children's Hospital, Vienna
- Belgium (7):
  - Antwerp University Hospital, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Regional De La Citadelle, Liège
  - CHC MontLegia, Liège
- Czechia (3):
  - University Hospital Brno, Brno
  - University Hospital Olomouc, Olomouc
  - Hospital Motol V Uvalu 841, Prague
- Denmark (3):
  - AUH Skejby, Aarhus
  - Copenhagen-Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Finland (4):
  - New Children's Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- France (16):
  - CHU Besancon, Besançon
  - CHU de Bordeaux, Bordeaux
  - HCE, Grenoble
  - CHRU de Lille, Lille
  - Institute of Hematology and Pediatric Oncology, Lyon
  - CHU Timone, Marseille
  - CHI Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU de Nice, Nice
  - Hôpital Robert Debré, APHP, Paris
  - TRS, Paris
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Charles Nicolle, Rouen
  - CHRU Strasbourg Hautepierre, Strasbourg
- Germany (16):
  - Universitätsklinikum Augsburg, Augsburg
  - Charite Universitaetsmedizin Berlin KöR, Berlin
  - Universitaetsklinikum Bonn AöR, Bonn
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitaetsklinikum Erlangen AöR, Erlangen
  - Justus-Liebig-Universitaet Giessen, Giessen
  - Universitaetsklinikum Halle (Saale) AöR, Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Universtitätsklinikum Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg AöR, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein AöR, Kiel
  - HELIOS Klinikum Krefeld GmbH, Krefeld
  - Johannes Gutenberg University Mainz, Mainz
  - Universitaetsklinikum Muenster AöR, Münster
  - Klinikum Der Landeshauptstadt Stuttgart gKAöR, Stuttgart
  - Universitaetsklinikum Tuebingen AöR, Tübingen
- Greece (4):
  - Aghia Sophia' Children's Hospital, Athens
  - HeSPHO, Athens
  - University General Hospital Of Heraklion, Heraklion
  - Mitera, Marousi
- Hungary (2):
  - University Semmelweis, Budapest
  - University of Pécs, Pécs
- National Children's Cancer Service, Dublin, Ireland
- Italy (4):
  - L'Azienda Ospedaliera Di Rilievo Nazionale Santobono-Pausilipon, Napoli
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma
  - Istituto Di Ricovero E Cura A Carattere Scientifico Materno Infantile Burlo Garofolo, Trieste
  - University Of Verona Medical School, Verona
- Japan (19):
  - Chiba University Hospital, Chiba
  - Ehime University Hospital, Ehime
  - Hiroshima University Hospital, Hiroshima
  - Hokkaido University Hospital, Hokkaido
  - Hyogo Prefectural Kobe Childrens Hospital, Hyōgo
  - Kagoshima University Hospital, Kagoshima
  - Kanagawa Childrens Medical Center, Kanagawa
  - Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Mie University Hospital, Mie
  - Nagoya University Graduate School of Medicine, Nagoya
  - Osaka City General Hospital, Osaka
  - Osaka University Graduate School of Medicine 2-2, Osaka
  - Saitama Prefectural Childrens Medical Center, Saitama
  - Shizuoka Childrens Hospital, Shizuoka
  - National Center for Child Health and Development, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Tokyo Metropolitan Childre's Medical Center, Tokyo
  - Tohoku University Hospital, Tōhoku
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Princess Máxima Center for pediatric oncology, Utrecht, Utrecht, Netherlands
- Christchurch Children's Hospital, Christchurch, New Zealand
- Norway (2):
  - Haukeland University Hospital, Bergen
  - St. Olavs Hospital, Trondheim
- Instituto Portugues de Oncologica Lisboa, Lisbon, Portugal
- Saudi Arabia (2):
  - Jeddah-King Abdulaziz Medical City, Jeddah
  - King Abdulaziz Medical City, King Abdullah International Medical Research Center, Riyadh
- National Institute of Children's Diseases, Bratislava, Slovakia
- Spain (4):
  - Vall D'hebron Institut De Recerca, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - University Hospital Virgen Del Rocio S.L., Seville
  - Hospital Universitario Y Politecnico La Fe, Valencia
- Sweden (6):
  - Childrens Cancer Center Queen Silvia Children´s Hospital, Sahlgrenska University Hospital, Gothenburg
  - Linkoping University Hospital, Linköping
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Umea University Hospital, Umeå
  - Children's UH, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in a publication
Supporting Information: CSR
Time Frame: The Clinical Study Report (CSR) will be made available within 6 months upon study end.
Access Criteria: A summary of the study results will be made public via www.clinical trials.gov as well as to Ethical committees/ Health Authorities and all participating patients by providing them through their treating physicians a patient letter with a summary of the results.